CLINICAL TRIAL: NCT02469025
Title: Effects of Grade III Traction-mobilization in End-range Joint Position in Patients With Hip Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Maria Fortun Agud, Unidad de Investigación en Fisioterapia, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI13/0030
Record Dates: First submitted 2015-05-26; First posted 2015-06-11 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Resting position mobilization group (Experimental): This group receive six manual therapy interventions based on manual traction mobilization in a resting position of the hip joint.
  In addition the physical therapist teach the patients six exercises to do at home between manual mobilization sessions.
  Interventions: Other: Manual caudal traction mobilization in resting position; Other: Selftreatment
- End range position mobilization group (Experimental): This group receive six manual therapy interventions based on manual traction mobilization in an end range position of the hip joint.
  In addition the physical therapist teach the patients six exercises to do at home between manual mobilization sessions.
  Interventions: Other: Manual caudal traction mobilization in end range position; Other: Selftreatment

INTERVENTIONS:
Other: Manual caudal traction mobilization in resting position
  Arms: Resting position mobilization group
Other: Manual caudal traction mobilization in end range position
  Arms: End range position mobilization group
Other: Selftreatment — Each subject is advice to do some exercises at home

SUMMARY:
Lower limb osteoarthritis is a major health problem in the westernized countries. The current gold standard treatment is joint replacement. However clinical guidelines recommend physical therapy as first option for these patients. Manual therapy has reported good reports in function, range of motion and pain in patients with hip osteoarthritis. The main aim of this study is to test the effects of a manual therapy protocol based on manual traction mobilization of the hip joint in an end range position and compare them with the effects achieve with the same protocol based on manual traction mobilization of the hip joint in a resting position. The investigators will use the caudal traction mobilization described by Kaltenborn. The study will test the effects of both treatments in passive range of motion, function and pain after three weeks of treatment, three weeks after finalizing the treatment and six weeks after.

ELIGIBILITY:
Inclusion Criteria:

* Hip osteoarthritis diagnosis
* Diminished range of motion
* Sign the informed consent

Exclusion Criteria:

* Contraindications to Manual Therapy.
* Sensitivity impairments in low back, pelvis, knee or foot regions.
* Being involved in other physical therapy treatments
* To change medication use during the study

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Passive Hip Range of Motion after intervention, at 3 weeks post-intervention and at 6 weeks post intervention | 3 weeks, 6 weeks, 9 weeks

SECONDARY OUTCOMES:
Changes from Baseline in Functional Tests (TUG, fast-paced walk test, stair climb test, 30sec. chair stand test), after intervention, at 3 weeks post-intervention and at 6 weeks post intervention | 3 weeks, 6 weeks, 9 weeks
Change from Baseline in Pain on the Visual Analog Scale after intervention, at 3 weeks post-intervention and at 6 weeks post intervention | 3 weeks, 6 weeks, 9 weeks
Change from Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale after intervention and at 6 weeks post intervention | 3 weeks, 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación en Fisioterapia. Universidad de Zaragoza, Zaragoza, Spain